CLINICAL TRIAL: NCT04648878
Title: A Comparison of Conventional Physical Therapy, Powered Exoskeleton, and Hybrid Physical Therapy With Exoskeleton in the Treatment of Individuals With Sub-acute and Chronic Stroke.
Brief Title: A Comparison of Conventional Physical Therapy, Powered Exoskeleton, and Hybrid Physical Therapy With Exoskeleton
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loma Linda University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 5190407
Record Dates: First submitted 2020-11-24; First posted 2020-12-02 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Stroke
Keywords: Stroke; Exoskeleton; Gait; Physical Therapy; Motor-learning
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Care Provider
Masking Description: participants will be instructed to not reveal which treatment arm they have been assigned to
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A - Hybrid combination (Experimental): Group A (n=12) will receive 18 alternating visits of conventional physical therapy and powered exoskeleton gait training with a wearable robotic powered exoskeleton , three times a week for approximately 6 weeks.
  Interventions: Other: Hybrid combination of physical therapy and powered exoskeleton
- Group B - Powered Exoskeleton only (Experimental): Group B (n=12) will receive 18 visits of powered exoskeleton only, three times a week for approximately 6 weeks.
  Interventions: Other: Powered Exoskeleton Only
- Group C - Physical Therapy only (Experimental): Group C (n=12) will receive 18 visits of physical therapy, three times a week for approximately 6 weeks. Upon completion of the data collection portion of the study, group C will receive 9 sessions, three times a week for approximately three weeks of powered exoskeleton therapy. Data will not be collected or reported during this phase, but but may be retained for future approved use.
  Interventions: Other: Physical Therapy only

INTERVENTIONS:
Other: Hybrid combination of physical therapy and powered exoskeleton — 18 alternating visits of conventional physical therapy and powered exoskeleton gait training with a wearable robotic powered exoskeleton , three times a week for approximately 6 weeks
  Arms: Group A - Hybrid combination
Other: Powered Exoskeleton Only — 18 visits of powered exoskelton only, three times a week for approximately 6 weeks
  Arms: Group B - Powered Exoskeleton only
Other: Physical Therapy only — 18 visits of physical therapy only, three times a week for approximately 6 weeks
  Arms: Group C - Physical Therapy only

SUMMARY:
The purpose of this investigator-initiated study is to establish if powered exoskeleton therapy as a part of a rehabilitation program can be used as a standard of care in stroke rehabilitation.

DETAILED DESCRIPTION:
This prospective randomized control trial with three treatment arms will begin by:

* Determining if the subject is a candidate for exoskeleton treatment.
* Randomly assigning subjects to three groups (physical therapy only, exoskeleton only, or a hybrid of physical therapy and exoskeleton).
* Body measurements to individualize the fit of the exoskeleton to each subject at each session.
* Activities-based balance confidence (ABC) questionnaire will be administered before and after the study begins.
* Timed up and go test (TUGT).
* Ten-meter walk test (10MWT).
* Six-minute walk test (6MWT)
* Berg Balance Test (BBT).
* Five times sit to stand (5XSTS).
* Heart rate through a portable heartrate monitor.

ELIGIBILITY:
Inclusion Criteria:

* Males and Females 18 years of age or older post-stroke

  * 3 Ashworth score are involved in a standing program less than 220 lbs 5'0" through 6'4" have the ability to follow one-step commands near normal range-of-motion for the knees, hips, and ankles

Exclusion Criteria:

* Exclusion criteria will include those who have already experienced powered exoskeleton therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2021-02-14 (Actual); Primary Completion 2024-11-20 (Actual); Study Completion 2024-12-18 (Actual)

PRIMARY OUTCOMES:
Timed up and go test | Pre and post tests up to six weeks apart
  Subject sits in a standard armchair and stands, and at a self-selected walking speed, walks 3 meters, turns, and walks back to the chair, and sits down. They will be timed. Takes three minutes to administer.
Ten meter walk test | Pre and post tests up to six weeks apart
  Subjects will be timed as they walk a known distance of 10 meters to determine his self-selected walking velocity (distance/time). They will be timed. Takes five minutes to administer.
6 minute walk test | Pre and post tests up to six weeks apart
  This test measures distance walked in six minutes to assess a patient's physical endurance. They walk at a self-selected speed and will be timed. This test takes approximately 10 minutes to administer
Berg Balance Test | Pre and post tests up to six weeks apart
  The Berg balance test is a reliable measure for predicting risk for fall. This 14-item test measures static and dynamic balance measures and takes 15-20 minutes to administer
The Activities-specific Balance Confidence (ABC) Scale | Pre and post tests up to six weeks apart
  This has been shown to be an effective tool for assessing the psychological impact of balance impairment and falls and measuring an individual's balance confidence. Using a Likert scale, this self-administered test evaluates a person's confidence in balance over various activities. This 16-question test takes 5 to 10 minutes to complete.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Davidson, MSE MPH, Principal Investigator — Loma Linda University O&P
Locations (1):
- Loma Linda University, Loma Linda, California, United States